CLINICAL TRIAL: NCT00512733
Title: Validation of Dietary Calcium Questionnaires Using Diet Records
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Dairy Council of California (Other)
Responsible Party: Sponsor
Other Study IDs: H9291-26992
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
Keywords: Healthy volunteers

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Dairy products continue to be an important source of calcium, providing over half the calcium intake for most individuals. Educational interventions promoting adequate calcium intake with tools estimating dietary calcium that can be easily utilized by consumers would be a valuable asset to promoting skeletal health. Validation of these tools against standard dietary assessment methods enhances their utility. The Dairy Council of California has developed two dietary calcium questionnaires, one electronic and one in print, using known dietary sources of calcium including frequency of consumption and portion size. For these questionnaires to be effective in clinical and research settings they must be a valid measurement of dietary calcium intake. To measure the validity of the dietary calcium questionnaires one hundred seventy three women will complete the two dietary calcium questionnaires and one 3-day food record. The dietary calcium questionnaires will be validated against this established method of dietary intake measurement. The objective of this study is to validate two dietary calcium questionnaires that can be used in clinical and research settings against an established method of dietary intake measurement. It is hypothesized that both dietary calcium questionnaires will be a valid measurement of dietary calcium intake in women.

DETAILED DESCRIPTION:
The Dairy Council of California has developed two dietary calcium questionnaires, one electronic and one in print, using known dietary sources of calcium including frequency of consumption and portion size. For these questionnaires to be effective in clinical and research settings they must be a valid measurement of dietary calcium intake. To measure the validity of the dietary calcium questionnaires one hundred seventy three women will complete the two dietary calcium questionnaires and one 3-day food record. The dietary calcium questionnaires will be validated against this established method of dietary intake measurement. The objective of this study is to validate two dietary calcium questionnaires that can be used in clinical and research settings against an established method of dietary intake measurement.

ELIGIBILITY:
Inclusion Criteria:

* Independently living women over the age of 19 in generally good health.

Exclusion Criteria:

* Inability to keep a diet record
* Active gastrointestinal disease that limits or restricts diet
* Inability to understand and provide informed consent.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2006-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Mean calcium intake | 3 days
  Participants' 3-day food records were mailed to the study and examined for completeness and legibility. Missing or unclear items were corrected by telephoning the participant. Food records were entered into Food Processor Plus software (ESHA Research, Salem, OR) to determine nutrient content. For food items that were not in the software's database, nutrient content was determined by examination of labels, contact with food manufacturers, search of the US Department of Agriculture nutrient database, or estimation from ingredient content by an RD.
  At the initial study visit, participants completed a written questionnaire and the online questionnaire. Calcium intake was calculated using a built-in calculator in the online questionnaire and by hand using the instructions in the booklet for the written questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Sellmeyer, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States